CLINICAL TRIAL: NCT06504667
Title: To Validate Point Mini User Needs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination of funding
Sponsor: Point Designs (Industry)
Collaborators: University of Colorado, Denver (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 445969; 4R44HD113485-02 (NIH)
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Amputation; Traumatic, Hand; Amputation, Congenital
MeSH Terms: conditions — Amputation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Prosthesis (Experimental): Patient is temporarily fit with Point Mini finger prosthetic system
  Interventions: Device: Point Mini

INTERVENTIONS:
Device: Point Mini — The Point Mini finger prosthetic system consists of 1-4 ratcheting mechanical digits and mounting brackets

SUMMARY:
The objective of the device feasibility study will be to validate the user needs of the Point Mini system. This study will be a single group intervention model where one group of 5 children with partial-hand upper limb loss will be asked to perform several tasks. Successful completion of a task results in a fulfilled user need. Failure to complete a task results in an unfulfilled user need.

ELIGIBILITY:
Inclusion Criteria:

* Partial hand loss with at least index and/or middle fingers loss at the MCP level
* Intact thumb with full range of motion
* Fluent in English
* Between the ages of 5 and 15 years

Exclusion Criteria:

* Patients with a residual limb that is unhealed from the amputation surgery
* Unhealed wounds
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
VAL-1 | Day 1 (8 hours)
  User wears Point Mini(s) for a entire session without discomfort (Pass/Fail)
VAL-2 | Day 1 (10 minutes)
  User flexes and extends the Point Mini(s) without using contralateral hand ten times (Pass/Fail)
VAL-3.1 | Day 1 (10 minutes)
  User lifts a 10-25 lb bag with Point Mini(s) depending on age (Pass/Fail)
VAL-3.2 | Day 1 (10 minutes)
  User grips a hammer with Point Mini(s) and makes indentations into the wood (Pass/Fail)
VAL-4 | Day 1 (10 minutes)
  User releases Point Mini(s) while performing an active grasp by pressing the dorsal button ten times sequentially (Pass/Fail)
VAL-5 | Day 1 (10 minutes)
  User positions Point Mini(s) into each of the locking positions without binding (Pass/Fail)
VAL-6 | Day 1 (10 minutes)
  User activates spring-back mechanism ten times without failure by using (1) contralateral hand, (2) tabletop, and (3) side or thigh (Pass/Fail)
VAL-7 | Day 1 (10 minutes)
  User grips a 5 lb cylindrical smooth object using Point Mini(s) for 10 seconds (Pass/Fail)
VAL-8 | Day 1 (10 minutes)
  User picks up 4 coins from a smooth tabletop within 30 seconds (Pass/Fail)
VAL-9 | Day 1 (8 hours)
  User performs VAL-1 through VAL-8 without Point Mini releasing from mounting system (Pass/Fail)

CONTACTS AND LOCATIONS:
Overall Officials: Levin Sliker, PhD, Principal Investigator — CEO, Point Designs
Locations (2):
- United States (2):
  - University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado
  - Point Designs, Lafayette, Colorado

IPD SHARING:
Plan to Share IPD: No